CLINICAL TRIAL: NCT07015229
Title: The Relationship of Pain Score Course and Analgesic Intervention Timing With Clinical Outcomes in the Postanesthetic Period After Septorhinoplasty
Brief Title: Septorhinoplasty and Pain Score Course
Status: Not yet recruiting | Type: Observational
Sponsor: Istinye University (Other)
Responsible Party: Principal Investigator, İlke Dolgun, assoc. prof., Haseki Training and Research Hospital
Other Study IDs: haseki pacu cevahir
Record Dates: First submitted 2025-06-03; First posted 2025-06-11 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Visual Analogue Scale

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: septorhinoplasty — To provide scientific contribution to more effective and timely pain management strategies in the postoperative period by evaluating the time-dependent course of pain scores and the effect of analgesic intervention timing on clinical outcomes in patients who underwent septorhinoplasty and who are followed in the postanesthetic care unit.

SUMMARY:
To provide scientific contribution to more effective and timely pain management strategies in the postoperative period by evaluating the time-dependent course of pain scores and the effect of analgesic intervention timing on clinical outcomes in patients who underwent septorhinoplasty and who are followed in the postanesthetic care unit.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years of age or older,
* Being in ASA I-III class,
* Having undergone septorhinoplasty surgery under general anesthesia under elective conditions,
* Being monitored for at least 30 minutes in postoperative,
* Being conscious and able to assess pain with VAS.

Exclusion Criteria:

* Patients who have undergone surgical procedures other than septorhinoplasty (e.g. laparoscopic, gynecological, orthopedic, etc.)
* Inability to assess pain due to impaired consciousness, agitation, or sedation in the postoperative period
* History of opioid derivatives or continuous analgesic use in the preoperative period
* Cognitive impairment, psychiatric disease at a level that prevents communication, severe visual or hearing impairment
* History of neurological or neuromuscular disease
* Having undergone revision septorhinoplasty or other revision surgery
* Patients with VAS≥4 during their follow-up in the postoperative,

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18-65 years with ASA 1-3 who underwent elective septorhinoplasty
Sampling Method: Non-Probability Sample
Enrollment: 78 (Estimated)
Dates: Start 2025-06-25 (Estimated); Primary Completion 2026-01-04 (Estimated); Study Completion 2026-01-20 (Estimated)

PRIMARY OUTCOMES:
visual analogue scale | 60 minutes
  0:no pain, 10:worst pain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Alshehri AA. Comparative Evaluation of Postoperative Pain Scores and Opioid Consumption in Septorhinoplasty After Administration of Single-Dose Preemptive Paracetamol and Ibuprofen: A Randomized Controlled Trial. Int Arch Otorhinolaryngol. 2023 Aug 4;27(3):e471-e477. doi: 10.1055/s-0042-1749386. eCollection 2023 Jul. PMID 37564463
- [Result] Perianez CAH, Castillo-Diaz MA, Barbosa MH, De Mattia AL. Pain Predictors in Patients in the Postanesthesia Care Unit. J Perianesth Nurs. 2024 Aug;39(4):652-658. doi: 10.1016/j.jopan.2023.11.010. Epub 2024 Feb 3. PMID 38310508